CLINICAL TRIAL: NCT04491968
Title: Mindfulness Oriented Recovery Enhancement for Chronic Pain and Opioid Relapse as an Adjunct to Methadone Treatment
Brief Title: Mindfulness Oriented Recovery Enhancement for Chronic Pain and Opioid Relapse
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rutgers, The State University of New Jersey (Other)
Collaborators: University of Utah (Other); National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Nina A. Cooperman, Psy. D., Associate Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro2019001687; R33AT010109 (NIH)
Record Dates: First submitted 2020-07-09; First posted 2020-07-30 (Actual); Results first posted 2025-03-10 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-02

CONDITIONS: Opioid Use; Chronic Pain
MeSH Terms: conditions — Chronic Pain | interventions — 2-methylcyclopentadienyl manganese tricarbonyl; Therapeutics

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled trial.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness Oriented Recovery Enhancement (Experimental): The Mindfulness Oriented Recovery Enhancement arm will participate in eight, weekly, two-hour group sessions.MORE sessions involve mindfulness training to prevent opioid relapse and reduce pain, cognitive reappraisal to decrease negative affect and regulate opioid craving, and savoring to augment natural reward processing and evoke positive emotion. Each session begins with a mindful breathing meditation, followed by a debriefing session. The therapist then debriefs participants' homework practice of using mindfulness, reappraisal, and savoring skills to cope with pain and enhance well-being in everyday life. During this debrief of the homework. Next, new psychoeducational material is introduced. Sessions culminate with an experiential exercise, and close with a brief mindful breathing meditation. Participants are asked to practice 15 minutes of mindfulness/reappraisal/savoring skills each day.
  Interventions: Behavioral: Mindfulness Oriented Recovery Enhancement
- Methadone Treatment as Usual (Other): In the methadone programs, clients typically come to the clinic regularly to get their methadone dose. Clients see their clinic substance abuse counselor for individual counseling, usually weekly at the beginning of treatment, with decreasing frequency if they remain abstinent and progress through treatment. Depending on clients' stage of MMT and success with remaining abstinent from drugs, they may be required to attend clinic treatment groups. Also, some clients may choose to go to voluntary counseling, educational, or support groups.
  Interventions: Other: Methadone Treatment as Usual

INTERVENTIONS:
Behavioral: Mindfulness Oriented Recovery Enhancement — MORE sessions involve mindfulness training to prevent opioid relapse and reduce pain, cognitive reappraisal to decrease negative affect and regulate opioid craving, and savoring to augment natural reward processing and evoke positive emotion. Each session begins with a mindful breathing meditation, followed by a debriefing session. The therapist then debriefs participants' homework practice of using mindfulness, reappraisal, and savoring skills to cope with pain and enhance well-being in everyday life. During this debrief of the homework. Next, new psychoeducational material is introduced. Sessions culminate with an experiential exercise, and close with a brief mindful breathing meditation. Participants are asked to practice 15 minutes of mindfulness/reappraisal/savoring skills each day.
  Other Names: MORE
  Arms: Mindfulness Oriented Recovery Enhancement
Other: Methadone Treatment as Usual — In the methadone programs, clients typically come to the clinic regularly to get their methadone dose. Clients see their clinic substance abuse counselor for individual counseling, usually weekly at the beginning of treatment, with decreasing frequency if they remain abstinent and progress through treatment. Depending on clients' stage of MMT and success with remaining abstinent from drugs, they may be required to attend clinic treatment groups. Also, some clients may choose to go to voluntary counseling, educational, or support groups.
  Other Names: MMT, Treatment as Usual, TAU
  Arms: Methadone Treatment as Usual

SUMMARY:
The objective of this study is to rigorously examine the impact of online MORE, delivered through video conference, on opioid use and chronic pain among individuals receiving methadone maintenance treatment (MMT). This study is a randomized controlled trial to test the efficacy of online MORE on opioid use and chronic pain immediately after treatment and 8-weeks post-treatment as compared to treatment as usual (TAU) among 154 individuals in MMT. Further, mediators (i.e., metacognitive awareness, negative emotion regulation, and natural reward processing) and moderators (i.e., gender, race, income, mental health, trauma, and MMT phase) of treatment response will be explored.

DETAILED DESCRIPTION:
This study is a 2-arm individually randomized controlled trial design in which outcomes of MMT patients randomized to MORE are compared to outcomes of those randomized to treatment as usual (TAU). In this study (N=154), the investigators will randomize MMT patients with chronic pain to MORE (n=77) or TAU (n=77). The purpose of this study is to determine MORE's efficacy for increasing opioid abstinence relative to TAU. Individuals with pain who are receiving MMT for an opioid use disorder (OUD) will be recruited from two methadone clinics in New Jersey.

Participants will be recruited through flyers posted in the clinics, being approached by research assistants in the waiting room of their usual methadone clinic, and referral by clinic staff. The number of individuals who contact the study staff through the flyers or referral and who are approached by study staff in the clinics will be tracked. Number of individuals who refuse study participation and who consent to the study will also be tracked. If an individual is interested in study participation, a trained research assistant will lead the individual through the informed consent process in a private space.

Since MORE is a closed group, the cohorts of 14 participants at each site will be randomized to TAU or MORE. Once 14 participants at a particular clinic are enrolled and randomized the MORE group will begin.

Participants randomized to the MORE condition will participate in eight, weekly, two-hour group sessions, co-led by a clinic and study counselor. Each session will contain 7 participants and take place remotely, by video conference. Attendance at each session and reasons for missing sessions will be recorded. Participants randomized to the control condition will continue receiving treatment as usual.

All study participants will partake in a total of three interviews lasting up to 90 minutes and occurring, remotely, at baseline, 8- and 16- weeks post-baseline by telephone or video conference. Each participant will also complete a urine or saliva drug screen at each assessment. All attempts to reach participants to schedule follow-up assessments will be tracked. Participants will also complete cognitive testing (for approx. 30-45 minutes) at baseline and 8-weeks and ecological momentary assessments (EMA) conducted via smartphones or tablets, which will be provided to each participant by study staff. EMA participation will require the participant to respond to twice-daily prompts in which they will be asked a series of brief questions regarding their current mood and exposure to opioid triggers. Additionally, subjects will be asked to initiate responses when they experience serious craving or relapse to opioid use. Each EMA assessment will last approximately 3-5 minutes.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* Age ≥18
* Currently on methadone
* Experiencing non-malignant pain for a duration of 3 months or longer.

Exclusion Criteria:

* Severe cognitive impairment or active psychosis
* Suicide risk
* Inability to attend the MORE group, if randomized to that arm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Actual)
Dates: Start 2020-08-13 (Actual); Primary Completion 2022-06-08 (Actual); Study Completion 2022-06-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nina Cooperman, PsyD, Principal Investigator — Rutgers Robert Wood Johnson Medical School
Locations (1):
- Rutgers Robert Wood Johnson Medical School, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Yes
Analyses of data generated from this project will be shared with the scientific community through publications in peer-reviewed journals and presentations at scientific meetings. The proposed research will include data from approximately 154 individuals in methadone maintenance treatment. The final dataset will include self-reported demographic and behavioral data from interviews with the subjects and laboratory data from urine or saliva specimens provided. Because we will be following study participants, we will be collecting identifying information. The final dataset will be stripped of identifiers prior to release for sharing.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning 3 months and ending 36 months after study publication.
Access Criteria: Data and associated documentation will be available to research community scientists only under a data-sharing agreement that provides for: (1) a commitment to using the data only for research purposes and not to identify any individual participant; (2) a commitment to securing the data using appropriate computer technology; and (3) a commitment to destroying or returning the data after analyses are completed.

REFERENCES:
- [Derived] Cooperman NA, Lu SE, Hanley AW, Puvananayagam T, Dooley-Budsock P, Kline A, Garland EL. Telehealth Mindfulness-Oriented Recovery Enhancement vs Usual Care in Individuals With Opioid Use Disorder and Pain: A Randomized Clinical Trial. JAMA Psychiatry. 2024 Apr 1;81(4):338-346. doi: 10.1001/jamapsychiatry.2023.5138. PMID 38061786

RESULTS

PARTICIPANT FLOW:
Groups:
- Mindfulness Oriented Recovery Enhancement: Participants in the MORE plus usual care group attended 8 weekly, 2-hour group sessions, remotely, through video conferencing. Participants were provided with a tablet and data plan to ensure access to the internet. MORE sessions involved mindfulness to strengthen self-regulation of drug use and reduce pain, reappraisal to regulate negative emotions and reduce craving by contemplating drug use consequences, and savoring to increase positive emotions and augment natural reward processing.Participants were taught to replace the reward obtained from drug use by self-generating natural reward via mindfulness and savoring. MORE also included techniques designed to mindfully honor the recovery process and promote reflection on the reasons for taking MOUD. Each session began with a mindful breathing meditation, followed by group processing of the meditation. Next, therapists debriefed participants' weekly homework practice of mindfulness, reappraisal, and savoring skills. These group processing efforts involved social-behavioral learning principles including positive reinforcement and shaping to maximize learning and motivation. Psychoeducational material and experiential exercises were then introduced, and participants were asked to practice 15 minutes of mindfulness/reappraisal/savoring skills daily.
- Methadone Treatment (MT) as Usual: In MT programs, patients take methadone daily and come to the clinic regularly to get their dose. However, at the time of the study, most participants received doses at home due to the COVID-19 pandemic. MT clinic individual and group therapy (neither involving mindfulness) was usually delivered through telehealth due to the COVID-19 pandemic.
Period: Overall Study
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Started | 77 | 77
Completed | 65 | 71
Not Completed | 12 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual | Total
Number analyzed (Participants) | 77 | 77 | 154
Age, Continuous [Mean (Standard Deviation); unit: years] | 49.2 (10.9) | 47.7 (11.3) | 48.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 33 | 33 | 66
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 66 | 66 | 132
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 29 | 33 | 62
  White | 38 | 42 | 80
  More than one race | 10 | 2 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 77 | 77 | 154
Completed less than high school [Count of Participants; unit: Participants] | 19 | 17 | 36
Unemployed [Count of Participants; unit: Participants] | 66 | 66 | 132
Used opioids in the past 30 days [Count of Participants; unit: Participants] | 44 | 40 | 84
Uses any drugs in the past 30 days [Count of Participants; unit: Participants] | 62 | 50 | 112
Number of years on methadone [Mean (Standard Deviation); unit: years] | 4.2 (4.7) | 3.1 (4.3) | 3.6 (4.6)
Depression [Mean (Standard Deviation); unit: units on a scale] — Depression was measured with Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D scale is a widely used valid and reliable measure that consists of 20 items with potential scores ranging from 0 to 60. A score above 16 on the CES-D indicates clinically significant symptoms of depression. Higher scores on the CES-D indicates greater depression.
  units on a scale | 22.5 (11.6) | 22.6 (11.0) | 22.6 (11.2)
Anxiety [Mean (Standard Deviation); unit: units on a scale] — Anxiety was measured with the Beck Anxiety Inventory (BAI). The BAI is also a widely used, reliable, and valid scale that consists of 21 items with potential scores ranging from 0 to 63. A score of 16 or higher indicates clinically significant symptoms of anxiety. A higher score on the BAI indicates greater anxiety.
  units on a scale | 25.5 (14.1) | 23.3 (15.4) | 24.4 (14.7)
Pain [Mean (Standard Deviation); unit: units on a scale] — Participants were asked "How intense is your pain right now?" on a scale from 0 ("no pain") to 10 ("very intense pain") during two daily prompts over 16-weeks through ecological momentary assessment.
  units on a scale | 5.1 (2.7) | 5.2 (2.5) | 5.2 (2.6)

OUTCOME MEASURES:

1. Primary Outcome: Drug Relapse Through 16-weeks.
Description: Drug use as measured by self-report through EMA, follow-back, or urine screen.
Time Frame: 16-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
Participants | 39 | 44
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Treatment (MT) as Usual; Test type: Superiority; p = .02, proportional hazard regression; Hazard Ratio (HR) = .58, 95% CI 2-sided [.37 to .90]

2. Primary Outcome: Methadone Treatment Drop Out Through 16-weeks.
Description: Methadone treatment drop out as measured by clinic report.
Time Frame: 16-weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
Participants | 10 | 17
Statistical Analysis 1: Comparison: Mindfulness Oriented Recovery Enhancement vs Methadone Treatment (MT) as Usual; Test type: Superiority; p = .04, proportional hazard regression; Hazard Ratio (HR) = .41, 95% CI 2-sided [.18 to .96]

3. Secondary Outcome: Number of Days of Any Drug Use
Description: A variable for number of days of drug use over 16 weeks were computed by counting the greatest number of days of drug use recorded through ecological momentary assessment, the Addiction Severity Index, or drug screen.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
days | 13.9 (16.9) | 21.7 (23.8)

4. Secondary Outcome: Number of Days of Opioid Use.
Description: Number of days of opioid use, other drug use, and any drug use over 16 weeks were computed by counting the greatest number of days of drug use recorded through ecological momentary assessment, Addiction Severity, Index, or drug screen.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
days | 7.9 (13.2) | 8.5 (14.8)

5. Secondary Outcome: Number of Days of Other Drug Use.
Description: Number of days of other drug use as measured by self-report through EMA or timeline follow-back and verified by urine or saliva drug screen.
Time Frame: 16-weeks
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
days | 9.8 (14.8) | 18.3 (23.0)

6. Secondary Outcome: Changes in Craving
Description: Change in craving ecological momentary rating on scale from 0 (e.g., no craving) to 6 (intense craving) to 10 (very strong craving) .
Time Frame: 16-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 73 | 72
units on a scale | -.49 (.30) | -.35 (.15)

7. Secondary Outcome: Changes in Pain.
Description: Participants were asked "How intense is your pain right now?" on a scale from 0 (no pain) to 10 (very intense pain) during 2 daily prompts over 16 weeks through ecological momentary assessment. Twice daily reports were averaged per week. Reduction in weekly pain average from baseline to 16 weeks was calculated and compared between groups.
Time Frame: 16-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 73 | 72
units on a scale | -.62 (.16) | -.25 (.13)

8. Secondary Outcome: Changes in Depression.
Description: Depression was measured with Center for Epidemiologic Studies Depression Scale (CES-D). The CES-D scale is a widely used valid and reliable measure that consists of 20 items with potential scores ranging from 0 to 60. A score above 16 on the CES-D indicates clinically significant symptoms of depression. Higher scores on the CES-D indicates greater depression.
Time Frame: 16-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
units on a scale | -3.68 (1.09) | -2.36 (1.06)

9. Secondary Outcome: Changes in Anxiety.
Description: Anxiety was measured with the Beck Anxiety Inventory (BAI). The BAI is also a widely used, reliable, and valid scale that consists of 21 items with potential scores ranging from 0 to 63. A score of 16 or higher indicates clinically significant symptoms of anxiety. A higher score on the BAI indicates greater anxiety.
Time Frame: 16-weeks
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
Number analyzed (Participants) | 77 | 77
units on a scale | -2.51 (2.47) | 1.31 (1.42)

ADVERSE EVENTS:
Time Frame: 16-weeks
Arm/Group | Mindfulness Oriented Recovery Enhancement | Methadone Treatment (MT) as Usual
All-Cause Mortality (participants affected / at risk) | 2/77 | 0/77
Serious Adverse Events (participants affected / at risk) | 0/77 | 0/77
Other Adverse Events (participants affected / at risk) | 0/77 | 0/77

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-02-02): https://cdn.clinicaltrials.gov/large-docs/68/NCT04491968/Prot_SAP_001.pdf
  • Informed Consent Form (2022-07-01): https://cdn.clinicaltrials.gov/large-docs/68/NCT04491968/ICF_002.pdf